CLINICAL TRIAL: NCT04422626
Title: Data Collection on the Application of Cytokine Adsorption Therapy on Patients With Acute Respiratory Failure Caused by COVID-19
Brief Title: Data Analysis of the Cytokine Adsorption Treatment on Coronavirus Disease-19 (COVID-19) Patients With Respiratory Failure
Acronym: CYTOAID
Status: Withdrawn | Type: Observational
Why Stopped: The human resources required to start enrollment were not available anymore.
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: 20802-5/2020/EÜIG
Record Dates: First submitted 2020-06-06; First posted 2020-06-09 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: SARS-CoV-2; COVID-19
Keywords: CytoSorb; COVID-19; acute respiratory failure; cytokine; Intensive care unit; Sars-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Three tubes (less than 25 ml) of blood and 2 ml of saliva will be collected to detect different antibodies, just in case if the physician already ordered blood test. Additional puncture won't be carried out.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill COVID-19 patients, who receive CytoSorb therapy: Patients in ICU due to critical COVID-19 infection, who receive early (within the first 24 hours, but no later than 48 hours after intubation) CytoSorb therapy on consultant's discretion.

SUMMARY:
Severe sepsis and septic shock are some of the leading causes of mortality in intensive care unit (ICU) admitted COVID-19 patients. The main cause of early mortality is the uncontrolled release of inflammatory mediators leading to cardiovascular failure. CytoSorb, a recently developed, highly biocompatible hemadsorption device has been tested, which can selectively remove inflammatory mediators from the circulation. This device is currently commercially available, and in Europe, it has been approved for clinical use. Based on experience to date, this adsorption technique may influence the immune function; removing inflammatory mediators from the blood may improve organ functions and even increase the chances of survival. CYTOAID is an observational, non-interventional study to assess the effectiveness of early cytokine adsorption therapy in critically ill patients who have been admitted to the ICU because of COVID-19 infection. Data on the applied therapy on COVID-19 patients in ICU will be collected and analyzed. The patient's examination and therapy will be applied according to the current regulations at the clinics and the current professional standards. The study does not require any additional examination or intervention.

DETAILED DESCRIPTION:
In the early phase of sepsis, the activation of innate immunity plays a significant role. Immune cells enhance the production of pro-inflammatory mediators. These pro-inflammatory mediators are responsible for the development of immune response and the intensification of the inflammatory processes. To counteract this, anti-inflammatory mediators limit and alleviate inflammation. Critically ill septic patients with higher levels of both anti- and proinflammatory mediators are at higher risk for death. The main cause for early mortality is the uncontrolled release of inflammatory mediators leading to cardiovascular failure, while in the late phase of the disease, secondary infections and the subsequent multiorgan failure dominate due to the exhaustion of the immune functions and the subsequent insufficient protective mechanisms. Therefore, it has been suggested that the outcomes of severe sepsis can be improved by attenuating the inflammatory processes. A recently developed, highly biocompatible hemadsorption device has been tested that can selectively remove inflammatory mediators from the circulation. This device is currently commercially available, and in Europe, it has been approved for clinical use. Based on experience to date, this adsorption technique may influence the immune function; removing inflammatory mediators from the blood may improve organ functions and even increase the chances of survival.

During the study, data will be collected exclusively; the application of CytoSorb therapy will be considered by the current physician always on an individual basis. Data will be recorded during hospitalization (using the documentations of the ICU) and immediately after discharge.

This study is suitable for recording every step of medical care from the diagnosis of SARS-CoV-2 infection. To investigate the biomarkers and the genetic background that potentially play a role in the infection, biological samples will be also collected - by already indicated interventions during standard care, i.e. without additional intervention.

This study aims to describe cytokine adsorption therapy (CytoSorb) in general and to detect its most important features. The study would also like to assess the safety and cost-effectiveness of the therapy, evaluate specific interventions required during the treatment, and to assess the outcomes of the disease. This study can provide important data and expand our knowledge about COVID-19 and its treatment, as well as improve the outcomes of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* confirmed COVID-19 infection
* ICU admission
* Mechanical ventilation due to COVID-19 pulmonary complications
* Moderate to severe acute respiratory distress syndrome (ARDS)
* CytoSorb therapy indicated by the attending medical team preferably within the first 24 hours, but no later than 48 hours after intubation
* Informed consent for data collection

Exclusion Criteria:

* Unlikely survival for 24 hours according to the attending physician
* Acute onset of hemato-oncological illness
* Patient already on ECMO
* Immunosuppression: on chronic systemic steroid therapy (>10 mg prednisolon/day); immunosuppressive agents (i.e.: methotrexate, azathioprine, cyclosporin, tacrolimus, cyclophosphamide)
* Patients with transplanted vital organs
* Thrombocytopenia (<20,000/uL)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to ICUs requiring mechanical ventilation with proven COVID-19 infection and treated with CytoSorb.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in the partial pressure of oxygen/fraction of inspired oxygen (PaO2/FiO2) ratio after CytoSorb therapy | 24 months
  Change in the PaO2/FiO2 ratio after CytoSorb therapy as compared to baseline

SECONDARY OUTCOMES:
Change in inflammatory biomarker levels during treatment | 24 months
  Change in white blood cell count and c-reactive protein levels during treatment compared to the baseline
change in organ function | 24 months
  measured by sequential organ failure assessment (SOFA/sub-SOFA) score during treatment assessed by the treating physician
length of stay in ICU | 24 months
  given in days, assessed by the treating physician
length of hospital stay | 24 months
  given in days, assessed by the treating physician
Duration of mechanical ventilation | 24 months
  given in days, assessed by the treating physician
Duration of vasopressor therapy | 24 months
  given in days, assessed by the treating physician
Duration of renal replacement therapy | 24 months
  given in days, assessed by the treating physician
Occurrence of critical illness polyneuropathy and/or myopathy | 24 months
  assessed by the treating physician
need for extracorporeal membrane oxygenation (ECMO) | 24 months
  Number of patients progressing to the need for ECMO assessed by the treating physician
cost calculation | 24 months
  The financial demand of the treatment of COVID-19 infection spent on each patient will be calculated by a healthcare economist after the trial is completed.
device-related adverse and serious adverse events | 24 months
  Number of patients with device-related adverse and serious adverse events assessed by the treating physician
In-hospital mortality | 24 months
  Number of patients, who died during their hospital stay, assessed by the treating physician

CONTACTS AND LOCATIONS:
Overall Officials: Péter Hegyi, MD, PhD, DSc, Study Chair — Insitute for Translational Medicine, University of Pécs, HU

IPD SHARING:
Plan to Share IPD: No